CLINICAL TRIAL: NCT00848510
Title: A Phase I, Open-label, Dose-escalation Study to Investigate the Safety, Tolerability, PD and PK of EMD 525797 Using DCE-MRI as a PK Measure of Response in Colorectal and Ovarian Cancer Patients With Liver Metastases After Failure of Standard Therapy
Brief Title: EMD 525797 in Colorectal and Ovarian Cancer Patients With Liver Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62242-003; 2008-001820-30 (EudraCT Number)
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Colorectal and Ovarian Cancer Patients With Liver Metastases
MeSH Terms: interventions — Abituzumab

ARMS (1):
- EMD 525797 (Experimental)
  Interventions: Biological: EMD 525797

INTERVENTIONS:
Biological: EMD 525797 — Abituzumab will be administered as an intravenous infusion for an hour at a dose of 250 milligram (mg) to 1500 mg at Weeks 1, 3 and 5. In case of clinical benefit (stable disease [SD], complete response [CR], or partial response [PR]) that will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST Version 1.0) during initial 6 Weeks, subjects will be allowed to continue treatment at the start of Week 7 at the given dose (250 mg or 500 mg or 1000 mg or 1500 mg) every second week until intolerance to treatment, withdrawal of consent, or the subject is no longer benefiting from treatment in the opinion of the Investigator.

SUMMARY:
This study is intended to test an experimental drug called EMD 525797 (Abituzumab). This drug is not yet approved for sale and has only been tested in a small number of people to date (prior to this study starting another research study was carried out involving 37 healthy volunteers receiving the study drug). Until more is known about this study drug, it can only be used in research studies.

This research study is planned to answer important questions about how the study drug is tolerated and how it may work in subjects with ovarian and colorectal cancer which has spread to the liver (i.e. metastatic cancer). The Sponsor (Merck KGaA) of this study is developing the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent
* Male or female subjects, aged at least 18 years
* Subjects with liver metastases (3 to 10 centimeter [cm] diameter) from colorectal and ovarian cancers
* Failure of standard cancer therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at study entry and an estimated life expectancy of at least 3 months
* Adequate haematological function, defined by absolute neutrophil count (ANC) greater than or equal to (>=) 1.5 x 10^9 per liter (/L), platelet count >= 100 x 10^9 / L, and haemoglobin concentration >= 9 gram per deciliter (g/dL)
* As subjects with documented liver metastases are treated in this trial, liver function test values are accepted as followed: up to the upper limit of Grade 2 as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0. This includes total bilirubin level less than or equal to (=<) 3 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels =<5 x ULN
* Adequate renal function defined by serum creatinine =<1.5 x ULN or a creatinine clearance of >=50 milliliter per minute (mL/min) calculated by Cockcroft-Gault
* Effective contraception (example: double barrier method) for both male and female subjects if the risk of conception exists. These subjects must be willing to avoid pregnancy during the study (screening to end of study [EOS]) as well as for at least 3 months after the last dosing.

Exclusion Criteria:

* Any systemic cancer treatment within 30 days before treatment with EMD 525797
* Thrombolytics or oral or parenteral anticoagulants (except to maintain patency of preexisting, permanent indwelling intravenous catheters) within 10 days prior to study start and during treatment
* Radiotherapy, chemotherapy, surgery, or any investigational drug in the 30 days before the start of treatment in this study, and/or diagnostic biopsies within 2 weeks before the start of treatment in this study
* Previous treatment with anti-integrin therapy or anti angiogenic therapy within the last 6 months
* Confirmed or clinically suspected brain metastases
* Known hypersensitivity reactions to the study medication
* History of allergic reactions to other monoclonal antibody (mAb) therapy
* Uncontrolled hypertension (systolic blood pressure greater than (>) 180 millimeter of mercury (mmHg), diastolic >100 mmHg)
* Current history of chronic daily aspirin therapy (doses of =< 150 mg is permitted), bleeding disorders, and/or history of thromboembolic events
* Severe peripheral vascular disease or ulceration
* Unstable angina pectoris, or myocardial infarction within 6 months before start of study treatment, clinical significant abnormal electrocardiogram (ECG) at screening;
* In women of childbearing potential, pregnancy (absence to be confirmed by beta human chorionic gonadotropin [β HCG] test, unless a subject has previously undergone hysterectomy or bilateral ovariectomy), or lactation period
* Known alcohol or drug abuse
* Participation in another clinical trial within the past 30 days before start of study treatment
* All other significant diseases which, in the opinion of the principal investigator (PI), might impair the subject's tolerance of study treatment
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Legal incapacity or limited legal capacity (not applicable only in rare cases)
* Known human immuno deficiency (HIV) infection and/or active hepatitis B or C virus infections
* Ongoing uncontrolled infections
* Contraindications to magnetic resonance imaging (MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Christie Hospital, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): Feb2009/Sep 2013. Study completion date: 28 Nov 2013. The study was conducted at 2 centers in United Kingdom and Spain.
Pre-assignment Details: Enrolled: 61 screened for eligibility; 20 excluded (mainly non-fulfillment of inclusion or exclusion criteria), 41 participants were enrolled into the study.
Groups:
- Abituzumab 250 mg: Abituzumab was administered as an intravenous infusion for an hour at a dose of 250 milligram (mg) at Weeks 1, 3 and 5. In case of clinical benefit (stable disease [SD], complete response [CR], or partial response [PR]) as assessed by the Response Evaluation Criteria in Solid Tumors version (RECIST) Version 1.0 during initial 6 Weeks, subjects were allowed to continue treatment at the start of Week 7 at the given dose every second week until intolerance to treatment, withdrawal of consent, or the subject was no longer benefiting from treatment in the opinion of the Investigator.
- Abituzumab 500 mg: Abituzumab was administered as an intravenous infusion for an hour at a dose of 500 mg at Weeks 1, 3 and 5. In case of clinical benefit (SD, CR, or PR) as assessed by the RECIST Version 1.0 during initial 6 Weeks, subjects were allowed to continue treatment at the start of Week 7 at the given dose every second week until intolerance to treatment, withdrawal of consent, or the subject was no longer benefiting from treatment in the opinion of the Investigator.
- Abituzumab 1000 mg: Abituzumab was administered as an intravenous infusion for an hour at a dose of 1000 mg at Weeks 1, 3 and 5. In case of clinical benefit (SD, CR, or PR) as assessed by the RECIST Version 1.0 during initial 6 Weeks, subjects were allowed to continue treatment at the start of Week 7 at the given dose every second week until intolerance to treatment, withdrawal of consent, or the subject was no longer benefiting from treatment in the opinion of the Investigator.
- Abituzumab 1500 mg: Abituzumab was administered as an intravenous infusion for an hour at a dose of 1500 mg at Weeks 1, 3 and 5. In case of clinical benefit (SD, CR, or PR) as assessed by the RECIST Version 1.0 during initial 6 Weeks, subjects were allowed to continue treatment at the start of Week 7 at the given dose every second week until intolerance to treatment, withdrawal of consent, or the subject was no longer benefiting from treatment in the opinion of the Investigator.
Period: Overall Study
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Started | 10 | 13 | 8 | 10
Completed | 10 | 13 | 8 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects analysis set included all subjects who entered the trial (that is, all subjects who signed informed consent).
Groups:
- Abituzumab 250 mg: Abituzumab was administered as an intravenous infusion for an hour at a dose of 250 mg at Weeks 1, 3 and 5. In case of clinical benefit (SD, CR, or PR) as assessed by the RECIST Version 1.0 during initial 6 Weeks, subjects were allowed to continue treatment at the start of Week 7 at the given dose every second week until intolerance to treatment, withdrawal of consent, or the subject was no longer benefiting from treatment in the opinion of the Investigator.
- Total: Total of all reporting groups
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg | Total
Number analyzed (Participants) | 10 | 13 | 8 | 10 | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (11.13) | 58.9 (9.94) | 68.9 (10.68) | 57.8 (16.58) | 61.2 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 3 | 8 | 22
  Male | 5 | 7 | 5 | 2 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Dose Limiting Toxicities (DLTs)
Description: Toxicity was graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. A DLT was defined as any Grade 3 or 4 haematological or non-haematological toxicity occurring during the first 4 weeks of treatment (that is, until the beginning of Week 5, with the exception of Grade 3 asymptomatic increase in liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], and alkaline phosphatase [ALP]) returning to Baseline within 7 days.), at any dose level, for which a causal relationship to the investigative medicinal product could not be ruled out by the Investigator and/or the Sponsor.
Time Frame: Up to Week 4
Population: Dose escalation analysis set included all subjects in the safety analysis set who experienced any DLT during the DLT observation period, regardless of the number of investigational medicinal product (IMP) administrations and subjects who received the IMP at Weeks 1, 3, and 5 for Cohort 1 and at Weeks 1 and 3 for all other cohorts.
Measure: Number; unit: Subjects
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 6 | 12 | 6 | 7
Subjects | 1 | 1 | 0 | 2

2. Primary Outcome: Volume Transfer Coefficient of Contrast Agent Across the Capillary Walls
Description: Volume transfer coefficient was defined as the volume transfer coefficient of contrast agent across the capillary wall, reflecting endothelial permeability and blood flow. Volumetric transfer coefficient was measured by dynamic contrast enhanced magnetic resonance imaging (DCE-MRI). DCE-MRI is a noninvasive quantitative method of investigating microvascular structure and function by tracking the pharmacokinetics of injected low molecular weight contrast agents as they pass through tumor vasculature.
Time Frame: Screening 1, screening 2, Week 1 Day 2, Week 1 Day 5, and Week 2 Day 1
Population: The DCE-MRI analysis set included all subjects who had at least one valid predose scan and at least one valid postdose (that is, after the infusion) scan.
Measure: Mean (Standard Deviation); unit: min^-1
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 8 | 12 | 8 | 10
min^-1
  Screening 1 | 0.233 (0.0817) | 0.214 (0.1385) | 0.221 (0.0991) | 0.141 (0.0650)
  Screening 2 | 0.253 (0.1219) | 0.177 (0.1450) | 0.176 (0.0851) | 0.137 (0.0602)
  Week 1 Day 2 | 0.227 (0.0869) | 0.175 (0.1048) | 0.180 (0.0769) | 0.136 (0.0676)
  Week 1 Day 5 | 0.227 (0.0934) | 0.165 (0.1154) | 0.171 (0.0665) | 0.132 (0.0723)
  Week 2 Day 1 | 0.209 (0.0992) | 0.171 (0.1039) | 0.194 (0.0938) | 0.156 (0.0687)

3. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation and TEAEs Leading to Death
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/ significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs were the AEs that occurred between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the initiation of the trial treatment until 30 days after last administration of trial treatment.
Population: The safety analysis set included all subjects who received at least one dose of IMP administration.
Measure: Number; unit: Subjects
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 10 | 13 | 8 | 10
Subjects
  TEAEs | 10 | 13 | 8 | 10
  Serious TEAEs | 5 | 7 | 5 | 7
  TEAEs leading to Discontinuation | 1 | 2 | 1 | 2
  TEAEs Leading to Death | 0 | 1 | 2 | 1

4. Secondary Outcome: Number of Subjects With Best Overall Response, Tumor Response and Clinical Benefit
Description: Tumor response was assessed by the Investigator, based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0 criteria. Tumor response was defined as the presence of a "best overall response" of complete response (CR) or partial response (PR). CR: Disappearance of all target and non-target lesions and/or normalization of serum levels of tumor markers. PR: At least a 30 percent decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of the LD of target lesions. The qualification of a CR or of a PR needed a confirmation by a second computed tomography (CT) scan at least 4 weeks after the first scan. Best overall response was derived programmatically as the best response recorded from the first investigation medicinal product administration until disease progression. Clinical benefit was defined as the presence of a "best overall response" of complete response or partial response or stable disease lasting at least 6 weeks.
Time Frame: Up to 4 years
Population: The full analysis set included all subjects who received at least one dose of IMP administration. "N" signifies the total number of participants evaluable for this outcome measure. Same subjects may be reported in more than one category.
Measure: Number; unit: Subjects
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 8 | 11 | 7 | 6
Subjects
  CR | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0
  SD | 0 | 2 | 1 | 0
  Progressive Disease | 8 | 9 | 6 | 5
  Not Assessable | 0 | 0 | 0 | 1
  Tumor Response | 0 | 0 | 0 | 0
  Clinical Benefit | 0 | 2 | 1 | 0

5. Secondary Outcome: Number of Subjects With Worsened Post Baseline Shift in ECOG Performance Status Score
Description: The number of subjects who experienced worse post baseline shift were assessed as per ECOG performance status score recorded during the treatment. The ECOG score is categorized as Grade 0, 1, 2, 3 and 4 where Grade 0=fully active, Grade 1=restricted in physically strenuous activity, Grade 2=unable to carry out any work activities, Grade 3=capable of only limited self-care and Grade 4=completely disabled.
Time Frame: Up to 4 weeks after last dose administration
Population: The safety analysis set included all subjects who received at least one dose of IMP administration.
Measure: Number; unit: Subjects
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 10 | 13 | 8 | 10
Subjects | 4 | 8 | 4 | 5

6. Secondary Outcome: Number of Subjects With Positive Binding Abituzumab Antibodies
Description: Subjects were defined as abituzumab positive if at least one positive result of antibodies against abituzumab was observed. In all other cases, subjects were defined as abituzumab negative.
Time Frame: Day 1 of Weeks 1, 3, 5, 6, 7, 8, and week 11 and end of study (EOS) visit (4 weeks after last dose administration)
Population: The immunogenicity analysis set included all subjects who received at least one dose of study drug administration and provided sufficient data from the antibodies samples. 'N' (number of subjects analyzed) signifies the subjects evaluable for this outcome measure. "n" signifies the number of subjects evaluable for each time point, respectively.
Measure: Number; unit: Subjects
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 9 | 11 | 7 | 7
Subjects
  Week 1 Day 1 (n=9,11,7,7) | 0 | 1 | 0 | 0
  Week 3 Day 1 (n=9,11,7,7) | 1 | 0 | 2 | 0
  Week 5 Day 1 (n=6,9,6,2) | 0 | 1 | 0 | 0
  Week 6 Day 1 (n=0,6,5,2) | 0 | 0 | 0 | 0
  Week 7 Day 1 (n=0,5,5,2) | 0 | 0 | 0 | 0
  Week 8 Day 1 (n=4,0,0,0) | 0 | 0 | 0 | 0
  Week 11 (n=0,1,3,0) | 0 | 0 | 0 | 0
  EOS Visit (n=6,3,2,1) | 1 | 0 | 0 | 0

7. Primary Outcome: Blood Plasma Volume and Extravascular/Extracellular Volume
Description: Blood plasma volume and extracellular/extravascular volume was measured using DCE-MRI.
Time Frame: Screening 1, screening 2, Week 1 Day 2, Week 1 Day 5, and Week 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 8 | 12 | 8 | 10
milliliter
  Blood Plasma Volume: Screening 1 | 0.024 (0.0162) | 0.014 (0.0071) | 0.020 (0.0122) | 0.022 (0.0183)
  Blood Plasma Volume: Screening 2 | 0.024 (0.0125) | 0.013 (0.0060) | 0.020 (0.0252) | 0.016 (0.0092)
  Blood Plasma Volume: Week 1 Day 2 | 0.019 (0.0078) | 0.014 (0.0090) | 0.015 (0.0114) | 0.020 (0.0191)
  Blood Plasma Volume: Week 1 Day 5 | 0.026 (0.0155) | 0.017 (0.0080) | 0.013 (0.0082) | 0.023 (0.0252)
  Blood Plasma Volume: Week 2 Day 1 | 0.028 (0.0201) | 0.019 (0.0087) | 0.019 (0.0220) | 0.020 (0.0164)
  Extravascular Volume: Screening 1 | 0.319 (0.0649) | 0.385 (0.1246) | 0.345 (0.1352) | 0.313 (0.0993)
  Extravascular Volume: Screening 2 | 0.302 (0.0559) | 0.319 (0.1007) | 0.307 (0.0860) | 0.307 (0.0808)
  Extravascular Volume: Week 1 Day 2 | 0.283 (0.0464) | 0.335 (0.1202) | 0.330 (0.0723) | 0.327 (0.0714)
  Extravascular Volume: Week 1 Day 5 | 0.271 (0.0531) | 0.327 (0.1162) | 0.336 (0.1080) | 0.312 (0.0924)
  Extravascular Volume: Week 2 Day 1 | 0.286 (0.0700) | 0.316 (0.1125) | 0.345 (0.0803) | 0.297 (0.0636)

8. Primary Outcome: Initial Area Under the DCE-MRI Contrast Agent Concentration Time Curve After 60 Seconds (IAUC60)
Description: IAUC 60 was used to give a gross indication of the delivery and uptake of contrast agent within the tumor (indicating the degree of perfusion and endothelial permeability. IAUC60 was measured using DCE-MRI.
Time Frame: Screening 1, screening 2, Week 1 Day 2, Week 1 Day 5, and Week 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: (Millimoles/liter)*sec
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 8 | 12 | 8 | 10
(Millimoles/liter)*sec
  Screening 1 | 21.900 (6.0987) | 20.844 (8.8439) | 22.752 (8.2156) | 16.602 (7.9627)
  Screening 2 | 21.155 (6.4053) | 17.670 (9.0159) | 19.437 (8.5201) | 16.168 (6.9961)
  Week 1 Day 2 | 22.513 (6.8728) | 18.140 (8.1305) | 18.724 (6.6599) | 17.607 (9.2052)
  Week 1 Day 5 | 21.006 (5.7951) | 17.557 (9.9606) | 18.758 (5.1517) | 16.313 (9.0325)
  Week 2 Day 1 | 20.356 (6.6613) | 18.498 (8.4957) | 20.201 (7.1768) | 17.314 (7.5539)

9. Primary Outcome: Whole Tumor Volume and Enhancing Tumor Volume
Description: Tumor volume (three-dimensional measurement) and the enhancing fraction of the tumor, which provides a gross measure of the proportion of the tumor that has a measurable level of perfusion, were assessed using DCE-MRI.
Time Frame: Screening 1, screening 2, Week 1 Day 2, Week 1 Day 5, and Week 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Cubic millimeter (mm^3)
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 8 | 12 | 8 | 10
Cubic millimeter (mm^3)
  Whole Tumor Volume: Screening 1 | 180310.380 (254443.5241) | 83921.304 (85983.0790) | 58662.341 (49075.1555) | 58665.247 (101041.3892)
  Whole tumor volume: Screening 2 | 195939.314 (268158.6384) | 73940.030 (81243.6227) | 57573.776 (48175.9173) | 63694.678 (121709.7593)
  Whole tumor volume: Week 1 Day 2 | 188556.463 (260719.8741) | 76214.685 (84401.6466) | 62941.056 (56871.6273) | 68159.203 (122487.7558)
  Whole tumor volume: Week 1 Day 5 | 195172.560 (264976.6619) | 72302.778 (79746.9479) | 68160.675 (61512.3298) | 74122.030 (135359.3601)
  Whole tumor volume: Week 2 Day 1 | 200316.632 (271342.9822) | 84412.235 (95360.1124) | 76755.877 (75170.5945) | 75468.633 (142025.4967)
  EnhancingTumor Volume: Screening 1 | 173882.006 (243514.1367) | 71043.485 (73510.7915) | 58160.983 (49084.1307) | 32790.886 (17602.3758)
  Enhancing tumor volume: Screening 2 | 190189.883 (259044.1496) | 70835.730 (75748.1887) | 56818.305 (48373.6133) | 68940.184 (118913.2150)
  Enhancing tumor volume: Week 1 Day 2 | 184552.465 (254423.3623) | 71323.352 (76071.6880) | 61519.396 (55375.5040) | 70147.221 (117332.7409)
  Enhancing tumor volume: Week 1 Day 5 | 189836.185 (256862.4972) | 71293.696 (75853.1409) | 66927.883 (61671.2327) | 74973.916 (133033.3585)
  Enhancing tumor volume: Week 2 Day 1 | 206074.402 (270622.8624) | 83616.930 (92140.5994) | 75835.576 (75420.1670) | 41201.278 (25012.0230)

10. Secondary Outcome: Progression-Free Survival (PFS) Time
Description: PFS was defined as the time from first study drug intake until radiological progression (based on RECIST Version 1.0) or death due to any cause. Only deaths within 84 days of last tumor assessment are considered. Subjects without event were censored on the date of last tumor assessment. Investigator read was the assessment of all imaging by the treating physician at the local trial site.
Time Frame: Time from first study drug intake to disease progression, death or last tumor assessment until end of trial visit (4 weeks after last dose administration)
Population: The safety analysis set included all subjects who received at least one dose of IMP administration.
Measure: Median (Full Range); unit: months
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Number analyzed (Participants) | 10 | 13 | 8 | 10
months | 1.22 [0 to 1.3] | 0.77 [0 to 7.6] | 1.40 [1 to 10.7] | 1.08 [0 to 1.2]

ADVERSE EVENTS:
Time Frame: From the initiation of the trial treatment until 30 days after last administration of trial treatment.
Arm/Group | Abituzumab 250 mg | Abituzumab 500 mg | Abituzumab 1000 mg | Abituzumab 1500 mg
Serious Adverse Events (participants affected / at risk) | 5/10 | 7/13 | 5/8 | 7/10
Other Adverse Events (participants affected / at risk) | 10/10 | 13/13 | 8/8 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abituzumab 250 mg (N=10) | Abituzumab 500 mg (N=13) | Abituzumab 1000 mg (N=8) | Abituzumab 1500 mg (N=10)
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 3
Asthenia (General disorders) | 0 | 1 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 2
Biliary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hepatobiliary infection (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abituzumab 250 mg (N=10) | Abituzumab 500 mg (N=13) | Abituzumab 1000 mg (N=8) | Abituzumab 1500 mg (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1
Hypochromic Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 2 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 4 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 4
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0 | 1
Asthenia' (General disorders) | 0 | 2 | 4 | 3
Early Satiety (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 2 | 1 | 5
Influenza like illness (General disorders) | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0
oedema peripheral (General disorders) | 1 | 2 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 2 | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1 | 3
Oral Herpes (Infections and infestations) | 1 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 2 | 1
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram Qt prolonged (Investigations) | 0 | 1 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 3 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 3 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 4 | 0 | 2
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Bladder Spasm (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 2 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis alergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 2 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other